CLINICAL TRIAL: NCT07128004
Title: Effect of Combined Acoustic Ripples and Transcranial Direct Current Stimulation on the Symptoms of New-Onset Subjective Tinnitus
Brief Title: In This Study, we Are Testing Whether Combining Two Interventions, in the Early Stages of Tinnitus, is More Effective in Quieting Tinnitus Than Using One Treatment Alone in the Later Stages of Tinnitus
Acronym: ATtDCS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Newcastle University (Other)
Collaborators: American Tinnitus Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: NU-019970; American Tinnitus Association (Other: American Tinnitus Association)
Record Dates: First submitted 2025-07-09; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Tinnitus; Acute
Keywords: Acute Tinnitus; Treatment; Sound therapy; tDCS
MeSH Terms: conditions — Tinnitus | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: principal researcher and participant are blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS and sound therapy active (Experimental): would present active tDCS and sound therapy for 40 minutes
  Interventions: Device: tDCS; Device: sound therapy
- tDCS and sound therapy sham (Sham Comparator): would provide a sham tDCS and sound therapy
  Interventions: Device: tDCS; Device: sound therapy

INTERVENTIONS:
Device: tDCS — would provide direct current for 40 minutes in 20 minute interval at 2 mA
  Other Names: transcranial direct current stimulation
Device: sound therapy — would provide acoustic ripples along with tDCS

SUMMARY:
* Tinnitus affects one in seven adults long-term
* Once present persistently for 4 weeks, tinnitus does not usually disappear
* People generally become less aware of, and less affected by, their tinnitus over time
* Only one in six people with tinnitus suffers a long-term negative impact on their life
* Current treatments can help to reduce the impact of tinnitus, but not silence the sound
* Treatments have only so far been tested once tinnitus has been present longer than 6 months
* In this study, the researchers are testing whether combining two interventions, in the early stages of tinnitus, is more effective in quieting tinnitus than using one treatment alone in the later stages of tinnitus
* One intervention (acoustic ripples) involves playing sounds through headphones for up to 60 minutes per day, and is mostly done in your own time
* The other intervention (transcranial direct current stimulation: tDCS) involves applying a weak electrical current to the volunteer's scalp using sponges soaked in salt water. This is performed in Newcastle University Medical School for a total of 8 sessions of 40 minutes each, spread over 4 weeks
* Half the volunteers will receive the 'real' intervention, and half a 'sham' or 'placebo' version. This will be randomly determined, and the volunteers or the research team will not known which you are receiving until the end of the study
* When the study ends, all volunteers will be able to use the 'real' intervention sounds in their own time, for as long as they wish, if they want to do so. No volunteers will be able to receive tDCS after the end of the study.
* All volunteers also complete questionnaires about their tinnitus, related symptoms and general health, and have hearing tests plus EEG (electrical brainwave) recordings
* The study is very low-risk, but does involve a total of 10 visits of around an hour each to Newcastle University Medical School over around a month. These can be arranged flexibly, including daytimes, evenings and weekends
* The researchers will pay all reasonable travel expenses, and £10 per hour for the volunteer's time in participating
* The study only completely ends 6 months after the date the tinnitus first started. At this point, the researchers will send some questionnaires to complete only. There is nothing to do for the study in between the tenth visit and this six-month questionnaire.

DETAILED DESCRIPTION:
Tinnitus is a common condition, in which people hear continuous sounds in the absence of an external source producing those sounds. Most people experience tinnitus for short periods of time throughout their life, for instance after exposure to loud noise, and some people experience long-term tinnitus. In most cases of tinnitus, there is a degree of hearing loss (often only mild), but it is rare for tinnitus to represent any serious disorder of the brain or ear. There are no widely effective treatments for tinnitus to reduce its loudness or eliminate it, but the majority of people with long-term tinnitus lead a normal life, without any impairment in quality of life on account of the tinnitus. A minority of people with long-term tinnitus experience distress as a result of it, and most people with long-term tinnitus gradually get used to the sound, and notice it less and less over time.

Previous studies have shown that applying a weak electrical current to the scalp (electrical stimulation) can lead to a small reduction in the loudness and impact of tinnitus for some people who have had tinnitus for many months or years already, and that this is significantly more effective, on average, than applying placebo (i.e. pretend) electrical stimulation. Electrical stimulation has never been tested in people who have recently developed their tinnitus.

Certain specific sounds, tailored to individuals' tinnitus, can significantly quieten tinnitus for some people, when these are listened to for an hour or so each day for weeks or months. However, the average quieting effect is quite modest. Like with electrical stimulation, these have only been tested by people with tinnitus already present for months to years.

Aims of study

The researchers believe that electrical stimulation and tailored sounds may be more effective in quieting tinnitus when given early in the course of tinnitus, compared to later on. Many researchers also believe that combining different types of tinnitus treatment may have a stronger effect than the sum of the effects of each individually.

Finally, the researchers want to test whether using interventions to quieten tinnitus early on in its course, even just for one month, might have a long-lasting or permanent effect in reducing tinnitus symptoms.

The benefits of treating tinnitus early, and using combination interventions, are currently theoretical, and one main aim of the study is to test whether they do exist.

The other main aim is to see how acceptable people find the course of combined intervention in the time period shortly after their tinnitus begins.

The volunteers are being approached because the volunteers have indicated that they have newly developed tinnitus.

What taking part involves

If they take part in the study, they will attend the researcher's laboratory on a total of 10 sessions over one month, to do the following:

* Provide details about their tinnitus and other health symptoms, and complete questionnaires (sessions 1 and 10 only)
* Undergo a hearing test (session 1 only). Note that this is not a substitute for having the volunteer's hearing formally assessed in a clinic.
* Undergo some computer-based sound tests (sessions 1 and 10 only). In these, they match a sound to the volume and pitch of their tinnitus so the researchers can estimate what it sounds like.
* Having an electroencephalography (EEG) recording, which measures their electrical 'brainwaves' (sessions 1 and 10 only)
* Have an electrical stimulation session for around 40 minutes (in each of sessions 2-9), which also includes listening to sounds through headphones.
* Provide quick symptom ratings of their tinnitus and its loudness before and after the electrical stimulation session. (sessions 2-9)

The first session may take up to 2 hours, and other sessions last around 1 hour each. The exact timing of the sessions can be negotiated with the research team to suit their schedule as far as possible. Weekday, evening and weekend appointments are all possible.

Separately to these sessions, we provide a copy of their personalised sound files to take home, and encourage you to listen to these for up to 60 minutes per day.

We will also contact them 6 months after the onset of their tinnitus to ask for them to report their current tinnitus symptoms, in the form of a questionnaire. This can be completed online, and does not require another visit.

ELIGIBILITY:
Inclusion Criteria:

* The presence of tinnitus (persistent sound heard in one or both ears that is not coming from an external sound source or actual sounds being generated inside your body such as turbulent blood flow), which has persisted for at least 3 days, and began within the last 8 weeks. You do not need to be aware of the tinnitus all the time, but it must be persistent in the sense that is can always hear it if you listen out for it, and there is not enough other sounds around to mask it.
* Age 18 or over
* The ability to make and communicate an informed choice about whether to take part in the study
* The ability to sit still and comfortably in a comfortable chair for around 1 hour at a time.

Exclusion Criteria:

* Tinnitus due to a physical sound source in the body, such as turbulent blood flow or muscle contractions in the middle ear.
* Presence of tinnitus over a period of 8 weeks
* Severe or profound hearing loss at high frequencies in the tinnitus ear(s), such that you could not properly hear the sounds used in the study
* Any implanted electronic device, such as a pacemaker, cochlear implant, bone-anchored hearing aid, nerve stimulator, deep brain stimulator or spinal cord stimulator
* Any areas of broken skin on the parts of the scalp where tDCS is applied
* Ménière's disease
* Any abnormality of brain structure (e.g. stroke, tumour), or other neurological disorder (e.g. multiple sclerosis or epilepsy)
* The ongoing use of sedating medications, or certain other nerve- or brain-acting medications
* A current mental health condition of sufficient severity to prevent certain activities of everyday life

In addition to these criteria, the researcher might have other reasons to suspect that participation is either contraindicated, or might be unsuitable. In such cases, the researcher should discuss these concerns with the potential participant and/or a senior member of the research team. Participation should only proceed if all those involved in these discussions agree it should.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-08-05 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-09 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Scale | 6 months for each participant
  Primary outcome will be perceived tinnitus loudness assessed using a self-reported Numerical Rating Scale (NRS), where participants rate the loudness of their tinnitus on a scale from 0 to 10. Higher scores indicate greater perceived loudness. The NRS will be administered at baseline and post-intervention to evaluate changes in subjective tinnitus loudness.

SECONDARY OUTCOMES:
Tinnitus Distress using Tinnitus Handicap Inventory | 6 months
  Tinnitus-related distress will be assessed using the Tinnitus Handicap Inventory (THI), a 25-item self-report questionnaire measuring the emotional, functional, and catastrophic impact of tinnitus. Higher scores indicate greater perceived handicap. The THI will be administered at baseline and post-intervention to evaluate changes in tinnitus-related distress.
Tinnitus distress using Tinnitus Functional Index | 6 months
  Tinnitus-related functional impact will be measured using the Tinnitus Functional Index (TFI), a validated 25-item questionnaire assessing tinnitus severity across eight subscales including sleep, emotional distress, and concentration. Higher scores reflect greater tinnitus-related burden. The TFI will be completed at baseline and post-intervention to assess changes in tinnitus-related impact.
Changes in tinnitus loudness | 6 months
  In addition to self-reported tinnitus distress, tinnitus loudness will be assessed using audiometric loudness matching, where participants adjust the intensity of a pure tone or narrowband noise presented to the ear ipsilateral to the tinnitus until it matches the perceived loudness of their tinnitus. The matched level will be recorded in decibels sensation level (dB SL), with measurements taken at baseline and post-intervention to evaluate changes in perceived loudness.

OTHER OUTCOMES:
Changes in source localized power and resting state functional connectivity | 6 months
  Exploratory measures will comprise resting-state electroencephalography (EEG) before and after the course of treatment, which will be analysed exploratively in terms of source-localised power and connectivity to indicate predictors of treatment success, correlates of treatment, and correlates of treatment success. 64-channel resting-state EEG data will be preprocessed in EEGlab, and transformed into source-level power and connectivity using the sLORETA toolbox. The following comparisons will be made using two-samples T tests or linear regression analyses with multiple comparisons correction:

CONTACTS AND LOCATIONS:
Overall Officials: William Sedley, PhD, Principal Investigator — Newcastle University

IPD SHARING:
Plan to Share IPD: Yes
Raw datas including participant's numerical rating scales, tinnitus questionnaires, and tinnitus pitch and loudness
Supporting Information: Study Protocol
Time Frame: Tentative from march 2027
Access Criteria: Access to raw data and study protocols

REFERENCES:
- [Background] Vanneste S, Byczynski G, Verplancke T, Ost J, Song JJ, De Ridder D. Switching tinnitus on or off: An initial investigation into the role of the pregenual and rostral to dorsal anterior cingulate cortices. Neuroimage. 2024 Aug 15;297:120713. doi: 10.1016/j.neuroimage.2024.120713. Epub 2024 Jun 27. PMID 38944171
- [Background] Umashankar A, Gander P, Alter K, Sedley W. Short- and long-term changes in auditory sensitivity and tinnitus distress between acute and chronic tinnitus: Longitudinal observation in a community-based sample. Hear Res. 2025 Jul;463:109299. doi: 10.1016/j.heares.2025.109299. Epub 2025 May 7. PMID 40378541

DOCUMENTS (1):
  • Study Protocol (2025-03-14): https://cdn.clinicaltrials.gov/large-docs/04/NCT07128004/Prot_000.pdf